CLINICAL TRIAL: NCT05742217
Title: MUltiple Myeloma Italian ObServational sTudy (MUST)
Brief Title: A Study to Learn How Patients With Triple Class Refractory Multiple Myeloma (TCR-MM) Are Treated in Italian Centers for Blood Related Diseases
Acronym: MUST
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071025; MUST (Other: Alias Study Number)
Record Dates: First submitted 2023-02-15; First posted 2023-02-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Multiple Myeloma (MM); Triple Class Refractory (TCR)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple myeloma (MM) is a type of cancer of the white blood cells, called plasma cells. These plasma cells help in fighting infections.

TCR-MM is when the cancer does not get treated with the 3 main classes of medicines used to treat this disease.

The purpose of this study is to learn about the present clinical practice in Italy and describe the standard of care that will be given to patients with TCR-MM, and their treatment costs, in around 25 centers who treat patients with blood diseases.

Standard of care (SoC) is the treatment that is accepted as a proper treatment for a certain type of disease and that is widely used by doctors.

The study is seeking for participants who are:

* 18 years of age or older
* Confirmed to have MM
* do not show any response when treated with the 3 main classes of medicines used to treat MM Data of participants who received the TCR treatment between 01 December 2021 and 31 May will be collected.

The main data source for the study will be the patient medical record. No clinical visits, examinations, or procedures are required as part of this study.

DETAILED DESCRIPTION:
In Italy, MM represents 1.6 percent of all cancers diagnosed in men and 1.5 percent of those diagnosed in women. The 2020 Italian epidemiological data show 5759 new diagnosis of MM. Most MM patients relapse or become refractory to various therapeutic approaches and typically cycle through many lines of treatment. Survival among patients refractory to newer therapies, including PIs, IMiDs and anti-CD38 mAbs, is very low and measured in months. An Italian real life data collection is important to analyse the current therapeutic approaches in TCR patients and the costs incurred by the therapy based on the different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of MM confirmed using International Myeloma Working Group (IMWG) criteria
* Patients are TCR defined as being refractory to all the 3 following classes: at least 1IMiD, at least 1PI and at least 1 anti-CD38 mA
* Relapsed/refractory to last anti-MM regimen prior to first treatment after TCR
* Started anti-MM treatment after TCR MM eligibility
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (at the date of first dose of first treatment after TCR MM eligibility, or no longer than 6 months prior to this date)
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study. Signed Patient informed consent and Privacy consent documents

Exclusion Criteria:

* Suffering from Smoldering MM
* Suffering from Plasma cell leukemia
* Suffering from amyloidosis
* Suffering from active Graft versus host disease (GvHD)
* Suffering from any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ
* Patients whose first treatment after becoming TCR was part of a clinical trial
* Participation in Elranatamab EAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have evidence of the following criteria in their medical records at the date of first dose of first treatment after TCR MM eligibility to be included in this study:
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Real-World Overall Response Rate (ORR) for each TCR MM therapy | 3-18 months
  The proportion of patients with confirmed Stringent Complete Response (sCR), Complete Response (CR), Very good partial response (VGPR), Partial Response (PR) by investigators per the International Myeloma Working Group (IMWG) criteria
Real-World Progression Free Survival (PFS) | 3-18 months
  The time from initiation of therapy until Progressive Disease (PD) by investigators per IMWG criteria or death due to any cause, whichever occurs first.
Real-World Overall Survival (OS) | 3-18 months
  Time from initiation of therapy until death due to any cause.
Real-World Duration of response (DOR) | 3-18 months
  For participants with an objective response (OR) per IMWG criteria, as the time from the first documentation of OR by investigators that is subsequently confirmed, until PD per IMWG criteria, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Italy (19):
  - A.O.U. - Ospedali Riuniti di Ancona, Torrette, Aviano
  - A.O.U. Policlinico S.Orsola Malpighi, Bologna, BO
  - "IRCCS "" Casa Sollievo della Sofferenza""tOpera di San Pio da Pietrelcina U.O.C di Ematologia", San Giovanni Rotondo, Foggia
  - AOU Policlinico Umberto I, Rome, Lazio
  - Fondazione IRCCS Policlinico Sa Matteo U.O.C. Ematologia, Pavia, Lombardy
  - A.O.U Policlinico G. Rodolico S. Marco, Catania, Sicily
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - A.O.O.R. Villa Sofia Cervello, U.O. Oncoematologia, Palermo, Sicily
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRST, Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola (FC)
  - A.O.U. Policlinico Università degli Studi di Napoli "Federico II", Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carita, Novara
  - Azienda Ospedaliero - Universitaria Di Parma, Parma
  - Ospedale Civile dello Spirito Santo, Pescara
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - AUSL della Romagna P.O. Ospedale Infermi U.O. di Oncologia, Rimini
  - Irccs Crob, Rionero in Vulture
  - San Giovanni Di Dio E Ruggi D'Aragona Hospital, Salerno
  - Busto Arsizio Hospital, Varese

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071025